CLINICAL TRIAL: NCT04838665
Title: Changes in Vital Signs and Pupil Diameter Related to Pharmacologic Mydriasis in Premature Infants: A Randomized Double Blind Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: OVS 2010-08-10-109
Record Dates: First submitted 2021-02-18; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Cyclopentolate; Phenylephrine; Tropicamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multiple Alternate Instillation of 0.5% cyclopentolate and 2.5% phenylephrine (MAI) (Active Comparator): 20 infants were enrolled in Multiple Alternate Instillation of 0.5% cyclopentolate and 2.5% phenylephrine (MAI)
  Interventions: Drug: 0.5% cyclopentolate and 2.5% phenylephrine; Drug: 0.5% tropicamide + 0.5% phenylephrine; Drug: 0.5% tropicamide + 0.5% phenylephrine with a cotton wick
- Single instillation of 0.5% tropicamide + 0.5% phenylephrine (SI) (Experimental): Single instillation of 0.5% tropicamide + 0.5% phenylephrine (SI)
  Interventions: Drug: 0.5% cyclopentolate and 2.5% phenylephrine; Drug: 0.5% tropicamide + 0.5% phenylephrine; Drug: 0.5% tropicamide + 0.5% phenylephrine with a cotton wick
- 1 instillation of 0.5% tropicamide +0.5% phenylephrine w/a cotton wick placed in the inferior fornix (Experimental): Single instillation of 0.5% tropicamide + 0.5% phenylephrine with a cotton wick placed in the inferior fornix (SIW)
  Interventions: Drug: 0.5% cyclopentolate and 2.5% phenylephrine; Drug: 0.5% tropicamide + 0.5% phenylephrine; Drug: 0.5% tropicamide + 0.5% phenylephrine with a cotton wick

INTERVENTIONS:
Drug: 0.5% cyclopentolate and 2.5% phenylephrine — Multiple Alternate Instillation of 0.5% cyclopentolate and 2.5% phenylephrine (MAI) dropped every 5 minutes for two doses
  Other Names: Multiple Alternate Instillation of Cyclopentolate Hydrochloride Dilate® Micro Labs Limited Bangalore and Phenylephrine Hydrochloride Mydfrin™ 25mg/mL (2.5%) Alcon Fort Worth Texas
Drug: 0.5% tropicamide + 0.5% phenylephrine — Single instillation of 0.5% tropicamide + 0.5% phenylephrine
  Other Names: Single instillation of Tropicamide + Phenylephrine Hydrochloride Sanmyd-P 0.5%/0.5% Santen Osaka Japan
Drug: 0.5% tropicamide + 0.5% phenylephrine with a cotton wick — Single instillation of 0.5% tropicamide + 0.5% phenylephrine with a cotton wick weighing 0.02 milligrams placed in the inferior fornix for the entire 45 minutes
  Other Names: Single instillation of Tropicamide + Phenylephrine Hydrochloride Sanmyd-P 0.5%/0.5% Santen Osaka Japan with a cotton wick placed in the inferior fornix weighing 0.02 milligrams

SUMMARY:
Retinopathy of prematurity (ROP) is one of the common anatomic causes of blindness among Filipinos, accounting for 47.7% of the cases. With this retinopathy being preventable and treatable, ROP screening has been proven to be effective in preventing blindness, which is achieved with the usage of mydriatics. Even if the regimen of multiple alternate instillations of 0.5% tropicamide and 2.5% phenylephrine is the one recommended by international guidelines for ROP screening, the mydriatic regimen used by many of the country's institutions is the single instillation of 0.5% tropicamide + 0.5% phenylephrine applied via a cotton wick placed in the inferior fornix (SIW). There have been no studies yet on the safety and efficacy in premature infants of this mydriatic preparation and method, although it is hypothesized that the usage of a cotton wick promotes the possible systemic effects of the mydriatic combination used.

This study then aims to determine the safety and efficacy of different mydriatic regimens in premature infants referred for screening of ROP using (1) multiple alternate instillations of 0.5% cyclopentolate hydrochloride and 2.5% phenylephrine (MAI), (2) single instillation of 0.5% tropicamide + 0.5% phenylephrine (SI), and (3) single instillation of 0.5% tropicamide + 0.5% phenylephrine with a cotton wick placed in the inferior fornix (SIW) in a tertiary Philippine hospital.

This study was designed as a randomized, double blind, clinical study which enrolled sixty preterm infants referred for ROP Screening from January to July 2011. With instillations via MAI, SI, and SIW, systolic blood pressure (SBP), diastolic pressure (DBP), mean arterial pressure (MAP), heart rate, and oxygen saturation were monitored from ten minutes prior to instillation up to forty-five minutes after instillation. Pupil dilations were also measured at the forty-fifth minute.

DETAILED DESCRIPTION:
I. Introduction Retinopathy of prematurity (ROP) is one of the common anatomic causes of blindness among Filipinos, accounting for 47.7% of the cases. With this retinopathy being preventable and treatable, ROP screening has been proven to be effective in preventing blindness, which is achieved with the usage of mydriatics. Even if the regimen of multiple alternate instillations of 0.5% tropicamide and 2.5% phenylephrine is the one recommended by international guidelines for ROP screening, the mydriatic regimen usually used by many of the country's institutions is the regimen of 0.5% tropicamide + 0.5% phenylephrine applied via a cotton wick placed in the inferior fornix. There have been no studies yet on the safety and efficacy in premature infants of this mydriatic preparation and method, although it is hypothesized that the usage of a cotton wick promotes the possible systemic effects of the mydriatic combination used.

II. Significance It is the aim of this study to evaluate the safety and efficacy of the mydriatic regimens we use in our institution and compare it to the recommendation by the UK ROP Guidelines. In doing so, this study aims to (1) document vital sign changes in the infant during dilation, (2) identify adverse systemic changes due to the mydriatic regimen and (3) provide appropriate interventions and recommendations to address these adverse effects. These will greatly improve the ROP screening process in our institution.

III. Objectives The general objective is to determine vital sign changes related to Pupil Dilation among preterm infants referred for ROP Screening from Neonatal Intensive Care Unit, Pediatric Wards and Eye Instrumentation Center of the Philippine General Hospital (PGH). Specifically, its objective is to compare the vital sign changes and mydriasis in (1) multiple alternate instillations of 0.5% Cyclopentolate Hydrochloride + 2.5% Phenylephrine (MAI) (2) single instillation of 0.5%/0.5% Phenylephrine + Tropicamide (SI) and (3) single instillation of 0.5%/0.5% Phenylephrine + Tropicamide with a cotton wick placed in the inferior fornix (SIW).

IV. Methodology This study was designed as a randomized, double blind, clinical study which enrolled sixty preterm infants referred for ROP Screening from January to July 2011. Each subject was randomly distributed into the standard, instillation, and packing group. To avoid observer bias, two investigators were involved per monitoring during dilation. The first investigator was assigned only to place the monitoring devices and to administer the mydriatics contained in unmarked 1 mL syringe which content was unknown to him.

The vital signs monitored during dilation were blood pressures (systolic, diastolic and mean arterial pressure (MAP)), heart rates and oxygen saturations using the newly calibrated Phillips Digital IntelliVue MP20 junior Cardiac monitors. A digital camera and a millimeter rule were used to approximate size of pupil dilatation. Measurement of all the vital signs and pupil dilation from a subject was derived from a single dilation session only.

Prior to data collection up to the end of monitoring, other factors that may affect the vital signs of the preterm infants were addressed. This included hunger, cold temperature, and soiled diapers.

Baseline vital signs determination was then performed 10 and 5 minutes prior to the first drop of mydriatic or proparacaine prior to packing. Additional reading will be done if there is a significant difference in the vital signs between 10 and 5 minutes prior to the initial drop.

For the MAI, multiple alternate drops of 0.5% cyclopentolate then 2.5% phenylephrine every 5 minutes in two doses were instilled (total of 0.2 milliliter of 0.5% cyclopentolate and 0.2 millimeter of 2.5% Phenylephrine). Vital signs were continuously recorded at time 0, 5, 10, 15, 20, 25, 30, 35, 40 and 45. At the 45th minute, a lid retractor was placed in the eyes of the subject after a drop of topical anesthesia. Pictures of the eyes were taken with a millimeter rule to serve as measurement reference.

For the SI, only a drop of 0.5%/0.5% tropicamide + phenylephrine was properly instilled at time 0 (total of 0.1 milliliter). Vital signs were continuously recorded at time 0, 5, 10, 15, 20, 25, 30, 35, 40 and 45. At the 45th minute, a lid retractor was placed in the eyes of the subject after a drop of topical anesthesia. Pictures of the eyes were taken with a millimeter rule to serve as measurement reference.

For the SIW, a cotton wisp soaked with a drop of 0.5%/0.5% tropicamide + phenylephrine was placed on the lower fornix in each eye of the infant (total of 0.1 milliliter). The weight of the cotton wisp was standardized at 0.02 milligram using a digital weighing scale. Vital signs were continuously recorded at time 0, 5, 10, 15, 20, 25, 30, 35, 40 and 45. At the 45th minute, a lid retractor is placed in the eyes of the subject after a drop of topical anesthesia. Pictures of the eyes were taken with a millimeter rule to serve as measurement reference. Pictures were uploaded into the computer monitor for the actual measurement.

Vital sign changes were monitored using the newly calibrated Phillips Digital IntelliVue MP20 junior Cardiac monitors. In the presence of significant vital sign changes, immediate intervention will be done.

In the presence of a significant increase in BP or heart rate, the infant will be observed. Both changes are expected from undergoing a stressful procedure such as placing a lid retractor in measuring the pupil dilation. The infant will be referred to the NICU ROD for further work up should tachycardia persist even after the examination. The blood pressure, heart rate and sensorium will be continuously monitored so as to avoid any ensuing bradycardia.

In the presence of a significant drop in BP, the infant will be referred to the NICU ROD for further work up to determine the possible source. Fluid challenge will be done to check if the cause of hypotension is just attributable to hypovolemia. The investigator will determine body temperature to check for hypothermia. If hypothermic, slow rewarming will be done by placing back the infant inside a close incubator or beside a radiant warmer. Blood glucose will be checked for hypoglycemia. Should hyperglycemia be detected, the infant can be started on 2cc/kg D5water. Infant will be worked up for infection as well.

During events of hypoxia or oxygen desaturation of less than 85%, the infant will be given supportive ventilation as required. Oxygen saturation will be monitored using the pulse oximeter. In the event of an apnea happening, supportive ventilation will be provided immediately, together with significant stimulation. The infant will be referred to the NICU ROD for possible intubation.

In the event of bradycardia, significant stimulation will be started on the infant. The infant will be referred to the NICU ROD for further work-up to determine the cause. The investigator is also to determine body temperature to check for hypothermia. If hypothermic, slow rewarming will be done by placing back the infant inside a close incubator or beside a radiant warmer. Blood glucose will be determined to check for hypoglycemia. Should hyperglycemia be detected, the infant can be started on 2cc/kg D5water. Infant can be worked up for infection as well.

In the event that a subject suffers from any of the abovementioned adverse effects, the appropriate interventions cited will be administered free of charge. Should the adverse effects believed by the investigators to be secondary to the ROP screening only and additional expenses are needed to procure medicines or equipment, the investigators will shoulder the expenses. If the medicine or equipment is immediately needed, the relative may spend first for them and have the expenses reimbursed with the investigators later. Should the amount to procure the said medicine or equipment cannot be produced by the relative, the investigators can be immediately contacted to assist the relatives immediately. All other expenses will be shouldered by the investigators through reimbursements. Expenses amounting to P500 for the medicine and P1000 for the equipment will be shouldered by the investigators. Should it exceed these limits, the infant will be referred to any charitable institution for further assistance.

The blood pressure (systole, diastole and MAP), HR and oxygen saturation obtained during dilatation were analyzed. They were graphed to determine patterns from baseline up to 45 minutes. Wilcoxon signed rank test was used to assess statistical significance for oxygen saturation, being a non-parametric variable. Poor dilatation among ROP patients with the advanced disease will be noted. A subgroup analysis was also done to determine the any relationship between the amounts of mydriatic used to the weight of the infant.

An interim analysis was done within the study to assess if the two mydriatic regimens were particularly beneficial or harmful compared to the concurrent standard group. Either the Pocock or the Flemming method will be used to decide if this study needed to terminate earlier than planned. Unblinding can be done should it be made necessary during the interim analysis or during course of the study. This protocol was submitted to the PGH ERB for ethics review and approval. It was conducted only upon approval from the ERB. All patient information were anonymized and are confidential. There is no funding received by the investigators for the conduct of this research.

ELIGIBILITY:
Inclusion criteria:

* birth weight of less than 1500 g
* gestational age of 32 weeks or less
* an unstable clinical course who are believed to be at high risk for Retinopathy of Prematurity, as assessed by their individual attendings

Exclusion criteria cited that

* infants with cardiac abnormalities directly affecting the heart rate and oxygen saturation
* infants with inotropic medications
* infants with ventilatory support

Ages: 1 Week to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure and systolic blood pressure changes | A baseline systolic blood pressure determination was performed 10 and 5 minute prior to the first drop of mydriatic or proparacaine prior to packing. Additional reading will be done if there is significant difference in the v/s between 10 and 5 minutes
  Measured in mmHg using a well-fitted neonatal cuff placed in the arm connected to the newly calibrated Phillips Digital IntelliVue MP20 junior Cardiac monitors
Diastolic blood pressure and diastolic blood pressure changes | A baseline diastolic blood pressure determination was performed 10 and 5 minutes prior to the first drop of mydriatic or proparacaine prior to packing. Additional reading will be done if there is significant difference in the vital signs between 10 and 5
  Measured in mmHg using a well-fitted neonatal cuff placed in the arm connected to the newly calibrated Phillips Digital IntelliVue MP20 junior Cardiac monitors
Mean arterial blood pressure and mean arterial blood pressure changes | A baseline mean arterial blood pressure determination was performed 10 and 5 mins. prior to the first drop of mydriatic or proparacaine prior to packing. Additional reading will be done if there is significant difference in the vital signs between 10 an
  Measured in mmHg using the newly calibrated Phillips Digital IntelliVue MP20 junior Cardiac monitors
Heart rate | A baseline heart rate determination was performed 10 and 5 minutes prior to the first drop of mydriatic or proparacaine prior to packing. Additional reading will be done if there is significant difference in the vital signs between 10 and 5 minutes prior
  Measured in beats per minute using the newly calibrated Phillips Digital IntelliVue MP20 junior Cardiac monitors
Oxygen saturation | A baseline heart rate determination was performed 10 and 5 minutes prior to the first drop of mydriatic or proparacaine prior to packing. Additional reading will be done if there is significant difference in the vital signs between 10 and 5 minutes prior
  Measured in percent saturation using a pulse oximeter connected to the newly calibrated Phillips Digital IntelliVue MP20 junior Cardiac monitors
Pupil diameter | Measured at the 45th minute post-instillation of the specified intervention
  Measuring using a digital camera and a millimeter ruler

SECONDARY OUTCOMES:
Successful retinopathy of prematurity screening | After the 45th minute measurement of pupil diameter
  Whether or not a successful ROP screening was carried out

CONTACTS AND LOCATIONS:
Overall Officials: Roland Joseph D Tan, MD, Principal Investigator — University of the Philippines Manila

IPD SHARING:
Plan to Share IPD: Undecided